CLINICAL TRIAL: NCT05084365
Title: A 6-month Study to Evaluate Sulforaphane Effects in Treatment of Cognition Impairment of PD Patients
Brief Title: A 6-month Study to Evaluate Sulforaphane Effects in PD Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD-Sulforaphane
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Sulforaphane; Parkinson's disease; cognition
MeSH Terms: conditions — Parkinson Disease | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sulforaphane (Experimental): The goal of the study is to investigate whether adding sulforaphane will benefit cognitive function in individuals who have PD.
  Interventions: Drug: Sulforaphane
- placebo (Placebo Comparator): The purpose of including placebo is to judge if the outcome is related to the study medication rather than other reasons.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulforaphane — Sulforaphane is a compound that can be extracted from broccoli, Brussel sprouts, cabbage, and other cruciferous plants.
  Arms: sulforaphane
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
Parkinson's disease (PD) is a second common neurodegenerative disease. More than 6 million individuals worldwide have Parkinson disease. No disease-modifying pharmacologic treatments are available. Current medical treatment is symptomatic, focused on improvement in motor (eg, tremor, rigidity, bradykinesia) and nonmotor (eg, constipation, cognition, mood, sleep) signs and symptoms. Accumulating evidence suggests the important role for inflammation and oxidative stress in the pathogenesis of PD. Sulforaphane extracted from broccoli sprout is an agent with potent anti-oxidant and anti-inflammatory activity. Previous studies suggested sulforaphane is useful in dopaminergic neuron survival. In this study, the investigator attempts to evaluate the efficacy and safety of sulforaphane in PD patients.

DETAILED DESCRIPTION:
The study will recruit 100 PD patients, and then these patients will be randomized to sulforaphane group or placebo group (50 patients per arm) for 24 weeks clinic trial. Participants will receive 24 weeks of either sulforaphane or placebo per day, in addition to the existing treatment. Baseline assessments include demographics, a comprehensive medical history, anthropometric measurements (weight and height), physical examination, and lab work. The motor symptoms and cognitive function will be assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) and MATRICS Consensus Cognitive Battery #MCCB#, respectively, at baseline, week 12 and week 24. The cranial MRI is examined at baseline and repeated at week 24. The primary outcomes will be the cognitive function improvement. Secondary outcomes include motor symptoms, biological data, MRI, safety and tolerability. During the study period, safety index including blood routine, liver and kidney function and adverse reactions report will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 40 to 75, regardless of ethnic group or gender;
2. Meeting the criteria for clinically established PD (2015) by Movement Disorder Association（MDS）; duration < 5 years;
3. Mini-Mental State Examination (MMSE) ≤ 27 points, but ≥20 points. Hoehn-Yahr stage ≤ 3;
4. Before enrollment, patients should take a stable dose of dopamine-based therapies drugs;
5. No obvious visual or hearing impairment;
6. More than 9 years of education;
7. Patients understand and comply with the study procedure, and are able to complete all tests and examinations required by the program. Sign the informed consent.

Exclusion Criteria:

1. Patients who have received globus pallidotomy, thalamotomy, deep brain stimulation (DBS), or stem cell therapy;
2. Other causes of parkinsonism: medications (e.g., metoclopramide, flunarizine), metabolic neurogenetic disorders (e.g., Wilson's disease), encephalitis, cerebrovascular diseases, or degenerative disorders (e.g., progressive supranuclear palsy);
3. Central nervous system diseases (including stroke, optic neuromyelitis, Parkinson's disease, epilepsy, etc.);
4. Have liver, kidney function insufficiency;
5. Unstable or severe diseases of the heart, lung, liver, kidney and hematopoietic system according to the judgment of the researchers;
6. Participated in other clinical trials within 3 months before screening visit;
7. Other conditions are unsuitable for participating in this study according to the judgement of researchers.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive improvement assessed using the MATRICS Consensus Cognitive Battery (MCCB) composite score | 24 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure.The MCCB total score is about 50 in healthy participants, the higher the score, the better the cognition performance.
Change of clinical symptoms by UPDRS | 24 weeks
  The change of UPDRS(Unified Parkinson Disease Rating Scale），ranging from 0-199, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, Principal Investigator — the Second Xiangya hospital, Central South University, 410011, Changsha, China.
Locations (1):
- Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided